CLINICAL TRIAL: NCT01767649
Title: Inflammatory Signature of Chorionic Cells as Markers of Premature Labor
Brief Title: Inflammatory Signature of Human Chorionic Cells
Acronym: TROPHY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI10056
Record Dates: First submitted 2013-01-11; First posted 2013-01-14 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Pregnancy
Keywords: Pregnancy; Remodelling; Extracellular matrix; Biomarkers
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood, placenta and maternal blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Caesarean: Normal pregnant women at term without complication during pregnancy and without inflammatory disorders
  Interventions: Other: Caesarean
- Vaginal Delivery: Normal pregnant women at term without complication during pregnancy and without inflammatory disorders
  Interventions: Other: Vaginal delivery

INTERVENTIONS:
Other: Caesarean — Collection of tissues and blood
  Groups: Caesarean
Other: Vaginal delivery — Collection of tissues and blood
  Groups: Vaginal Delivery

SUMMARY:
The purpose of this study is to identify molecules produced specifically by the cells from the chorionic membranes of the materno-fetal interface ("the water bag") sign for the activation of preterm labor.

DETAILED DESCRIPTION:
· Background

During human gestation, fetal membranes (the "water bag") encompass the amnion, facing the amniotic cavity, and the chorion, lining the maternal decidua and comprising trophoblast cells. Membranes usually remain intact until their spontaneous rupture, close to the first stage of labor at term. Often seen as a simple inert shell, with a role of "airbag" for the developing fetus, the membranes provide yet a large surface of interaction between maternal and fetal tissues and function as a transient endocrine organ with immune properties. Indeed human parturition is tightly correlated with hormonal changes at the maternal-fetal interface during pregnancy, that may control cell interactions and chorio-decidua remodeling, the amnion remaining usually intact until the final break. Precocious remodeling may lead to a premature onset of labor, associated or not with premature rupture of membrane whether the cause is infectious or not. A better understanding of this membrane remodeling may thus offer new avenues to define biomarkers of preterm labor.

Hereof, the fact that the mother-to-be accepts and keeps the fetus for months within her womb has long being seen as an enigma, since the fetus is a semi-allograft, half of his genome being of paternal, thus of foreign, origin. This apparent paradox was deciphered by the demonstration of the set-up of an immunotolerance at the site of implantation through the education of maternal immune cells (Natural Killer and T cells) by the fetal trophoblast. This immunotolerance is normally maintained throughout pregnancy, and some recurrent spontaneous miscarriages have been shown to be due to the loss of this immunotolerance, which activates the rejection of the semi-allograft.

In this regard, remodeled fetal membranes overlying the cervix may discharge signals that could be detectable in cervicovaginal fluids and serve as biomarkers of the imminence of delivery. Such information on delivery timing may be of great importance for an adequate prediction that would change drastically the management of threatening preterm delivery.

· Current proposal The objective of this study is to characterize the fetal and maternal cells in the chorio-decidua during the remodeling of the membranes using our well-established cell model (Hervé et al. 2008, J Immunol).

ELIGIBILITY:
Inclusion Criteria:

* >18y old
* Singleton
* Normal pregnancy without complication
* >37 weeks of gestation

Exclusion Criteria:

* Minor
* Without Health Insurance
* Inflammatory Disorders (diabetes, twin, autoimmune disesses, etc)
* Infection HIV, hepatitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal pregnant women followed for their pregnancy in the maternity
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Protein overexpression | 1 year
  Setting of measurements of proteins in the supernatant of chorionic cells

CONTACTS AND LOCATIONS:
Overall Officials: Céline Méhats, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- INSERM, Paris, France

REFERENCES:
- [Background] Herve R, Schmitz T, Evain-Brion D, Cabrol D, Leroy MJ, Mehats C. The PDE4 inhibitor rolipram prevents NF-kappaB binding activity and proinflammatory cytokine release in human chorionic cells. J Immunol. 2008 Aug 1;181(3):2196-202. doi: 10.4049/jimmunol.181.3.2196. PMID 18641359
- [Background] Mehats C, Schmitz T, Marcellin L, Breuiller-Fouche M. [Biochemistry of fetal membranes rupture]. Gynecol Obstet Fertil. 2011 Jun;39(6):365-9. doi: 10.1016/j.gyobfe.2011.04.006. Epub 2011 May 24. French. PMID 21602079